CLINICAL TRIAL: NCT06864806
Title: Development of a Protocol for Non-Invasive Prenatal Analysis of Cell-Free Circulating Fetal DNA (ccfDNA) Using Massively Parallel Sequencing (MPS)
Brief Title: Prenatal Analysis of Cell-free Circulating Fetal DNA
Acronym: APAFLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/80
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related
Keywords: Non-invasive; Prenatal analysis; ccfDNA; MPS; Paternal filiation; Sexual assault
MeSH Terms: interventions — Genetic Profile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic profile (Experimental): Filiation analysis between the fetus and his father
  Interventions: Other: Genetic profile

INTERVENTIONS:
Other: Genetic profile — Filiation analysis between the fetus and his father

SUMMARY:
In criminal cases involving sexual assault, victims may later discover they are pregnant, creating profound uncertainty about the paternity of the fetus. These distressing situations compound the trauma already experienced by the victims. To address this, the Medico-Legal Hematology Laboratory (LHML) in Bordeaux aims to validate a method based on Massively Parallel Sequencing (MPS) and a specific isolation protocol for analyzing cell-free circulating fetal DNA (ccfDNA) in maternal blood samples. This identification process will confirm or exclude paternal genetic relationships between the fetus and potential fathers between 6 and 22 weeks of amenorrhea. These analyses will only be conducted under judicial requisition, in accordance with the French Code of Criminal Procedure

DETAILED DESCRIPTION:
The objective of this study is to validate a non-invasive protocol for extracting and purifying ccfDNA from maternal blood samples and analyzing fetal DNA using MPS technology to establish paternity. To develop this methodology, a preliminary study will be conducted using blood samples from pregnant women whose partners' identities are known. LHML has partnered with Professor Sentilhes' team at Bordeaux University Hospital Center to obtain these samples.

Venous blood samples (~10 mL) will be collected from pregnant women between 6 and 22 weeks of amenorrhea in PAXgene Blood ccfDNA tubes (Qiagen) to prevent DNA degradation. The samples will be centrifuged to separate plasma, and ccfDNA will be isolated using the EZ2 Connect Fx instrument and the EZ1&2 ccfDNA kit (Qiagen). In parallel, buccal swabs will be collected from the mothers and their partners as reference samples, processed using LHML's routine DNA extraction protocols. Additionally, umbilical cord blood from newborns will be collected and processed with an in-house protocol to obtain purified DNA extracts.

These reference samples will allow us to confirm the profiles previously identified for the pregnant women and the fetuses but also to validate the filiation analysis between the fetus and his father. All DNA samples will be quantified using the Investigator QuantiPlex Pro kit (Qiagen) and the QuantStudio 5 Real-Time PCR System (Applied Biosystems).

ccfDNA from maternal blood will be analyzed using the MiSeq FGx Sequencing System (Verogen), the first NGS instrument validated for forensic genomics. The Verogen ForenSeq MainstAY Kit, which amplifies and sequences 27 autosomal STRs, 25 Y-STRs, and Amelogenin, will be used. This approach ensures reliable profiling even from low concentrated ccfDNA samples, with capacity for up to 96 libraries per run.

Reference DNA from buccal swabs and umbilical blood will undergo MPS using the same Verogen ForenSeq MainstAY Kit and be cross-validated with capillary electrophoresis using the Investigator 24Plex QS kit (Qiagen). Data analysis will be performed with the ForenSeq Universal Analysis Software and an in-house parentage analysis program developed by LHML. The Familias software may also be used to calculate likelihood ratios for paternity determination. All data processing systems are offline to ensure confidentiality.

This open prospective study will require samples from 20 complete triads (mother, father, newborn) and will address two major critical points. The first objective is to determine the quality threshold of the genetic profiles obtained with the Verogen ForenSeq MainstAY kit necessary for reliable paternity analysis. This will be assessed by calculating the percentage of validated STR loci among the 27 autosomal STRs analyzed. The second focus is to establish the optimal ccfDNA quantity required to generate a genetic profile covering at least 20 autosomal STRs using the Verogen ForenSeq MainstAY kit. This will involve quantifying the ccfDNA extracts and correlating these values with the maternal blood volume needed to obtain sufficient ccfDNA for analysis. Ultimately, this study aims to advance scientific understanding of ccfDNA analysis in pregnant women using MPS technology and, most importantly, to provide critical support to women who become pregnant following sexual assault by enabling them to confirm the paternity of their fetus with certainty, addressing a crucial aspect of their psychological recovery

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* For woman: pregnancy between 6 and 22 weeks
* For both mother and father: non-opposition to participate and genetic signed informed consent

Exclusion Criteria:

* Unknown paternity.
* Maternal blood-borne infections (HIV, syphilis, hepatitis B).
* Inability of the father to provide a sample.
* Insufficient comprehension of French by either parent.
* Mother or father under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Genetic profile | Baseline
  The quality of the genetic profile obtained with the ForenSeq MainstAY kit will be estimated as a percentage of validated markers (loci) among the 27 autosomal markers analyzed by the kit

SECONDARY OUTCOMES:
Free circulating fetal DNA | Baseline
  The quantity of circulating cell-free fetal DNA necessary for the establishment of a genetic profile will be measured from a minimum of 20 autosomal markers using the ForenSeq MainstAY kit This value will be measured by the concentration in ng/µl.
Maternal blood | Baseline
  Quantity of maternal blood necessary to obtain a sufficient quantity of circulating cell-free fetal DNA for genetic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France